CLINICAL TRIAL: NCT04898478
Title: Intervention Development and Pilot Study to Prevent Untreated Native Hawaiian and Pacific Islander Opioid Use Disorder
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, Riverside (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: R34DA049989 (NIH)
Record Dates: First submitted 2021-04-13; First posted 2021-05-24 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-04

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Seeking Intervention for Pacific Islanders with Opioid Use Disorders (Experimental): This arm will consist of a behavioral intervention to increase treatment seeking among Pacific Islanders with opioid use disorders.
  Interventions: Behavioral: Treatment Seeking Intervention for Pacific Islanders with Opioid Use Disorders

INTERVENTIONS:
Behavioral: Treatment Seeking Intervention for Pacific Islanders with Opioid Use Disorders — The investigators will design a culturally grounded treatment seeking intervention for Pacific Islanders with OUDs

SUMMARY:
This study will design and pilot/feasibility test a culturally grounded intervention to increase the treatment seeking of Pacific Islanders with opioid use disorders in formal services.

DETAILED DESCRIPTION:
For the clinical trial arm of this pilot/feasibility study, the investigators will conduct a pilot/feasibility test of our conceptual model of culturally grounded intervention components with 20 Pacific Islander adults with experience with opioid use disorders, then conduct 2 focus groups per site to finalize the components and items for larger R01 pilot and randomized wait-list controlled testing.

ELIGIBILITY:
Inclusion Criteria:

* Of Pacific Islander/Native Hawaiian or part-Pacific Islander/Native Hawaiian heritage.
* Live in Utah or Hawaii.
* For all lay Pacific Islander adult participants: must be over 18 years of age.
* Fluent (oral and reading) in English or Native Hawaiian.

For target Pacific Islander participants with OUDs, additional inclusion criteria is:

- Presence of active OUD, as screened via 8-item Rapid Opioid Dependence Scale.

Exclusion Criteria:

* Do not meet inclusion criteria,
* Are unwilling to participate,
* Fails to provide or retracts consent,
* Reside outside the target communities of Utah or Hawaii

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Pacific Islander Knowledge Scale about Opioid Use Disorders and Treatment | Up to 12 months
  5-point scale designed by the team to assess Pacific Islander knowledge of opioid use disorder and treatment with items such as "What causes most OUDs? What are the different treatment options for PIs with OUDs"

SECONDARY OUTCOMES:
Pacific Islander Attitude Scale about Opioid Use Disorders and Treatment | Up to 12 months
  10-point scale designed by the team to assess Pacific Islander attitudes toward opioid use disorder treatment such as "How important is treatment?" and "How scary is treatment?"

CONTACTS AND LOCATIONS:
Locations (1):
- UC Riverside, Riverside, California, United States

IPD SHARING:
Plan to Share IPD: Undecided